CLINICAL TRIAL: NCT00275756
Title: Effects of Common Topical Glaucoma Therapy on Optic Nerve Head Blood Flow Autoregulation During Increased Arterial Blood Pressure and Artificially Elevated Intraocular Pressure in Healthy Humans
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Gabriele Fuchsjaeger-Mayrl, MD, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: OPHT-040106
Record Dates: First submitted 2006-01-11; First posted 2006-01-12 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Glaucoma
Keywords: Ocular Physiology; Brimonidine; Timoptic; Dorzolamide; ocular blood flow; Regional Blood Flow
MeSH Terms: conditions — Glaucoma | interventions — Timolol; Pharmaceutical Preparations; dorzolamide; Brimonidine Tartrate; Laser-Doppler Flowmetry

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Timolol (drug); Device: Laser Doppler flowmetry; Device: Goldmann applanation tonometer; Procedure: Suction cup method
- 2 (Experimental)
  Interventions: Drug: dorzolamide (drug); Device: Laser Doppler flowmetry; Device: Goldmann applanation tonometer; Procedure: Suction cup method
- 3 (Experimental)
  Interventions: Drug: brimonidine (drug); Device: Laser Doppler flowmetry; Device: Goldmann applanation tonometer; Procedure: Suction cup method

INTERVENTIONS:
Drug: Timolol (drug) — Timolol (0.5%, non-selective beta-blocker, Timoptic®, Merck Sharp & Dohme, Haarlem, Netherlands), dose 1 drop in one eye twice daily for two weeks
  Arms: 1
Drug: dorzolamide (drug) — Dorzolamide (2%, carbonic anhydrase inhibitor, Trusopt®, Laboratoires Merck Sharp & Dohme - Chibret, France), dose: 1 drop in one eye twice daily for two weeks
  Arms: 2
Drug: brimonidine (drug) — Brimonidine (0.2%. alpha-2 adrenergic agonist, Alphagan®, Allergan Pharmaceuticals, Westport, Ireland), dose: 1 drop in one eye twice daily for two weeks
  Arms: 3
Device: Laser Doppler flowmetry — blood flow measurements at the temporal neuroretinal rim of the optic nerve head, in total 4x 9 minutes on 2 study days
Device: Goldmann applanation tonometer — intraocular pressure measurements, in total 2x 5 measurements on two study days
Procedure: Suction cup method — The IOP will be raised by an 11 mm diameter, standardized suction cup placed on the temporal sclera with the anterior edge at least 1 mm from the limbus; 4x 8 minutes on 2 study days

SUMMARY:
Background

Autoregulation is the ability of a vascular bed to maintain blood flow despite changes in perfusion pressure. The existence of an effective autoregulation in the optic nerve circulation has been shown in animals and humans. The exact mechanism behind this autoregulation is still unknown. The motive for the investigation of optic nerve head (ONH) blood flow autoregulation is to enhance the understanding of pathologic eye conditions associated with ocular vascular disorders. To clarify the regulatory mechanisms of ONH microcirculation is of critical importance to understand the pathophysiology of glaucoma, because there is evidence that glaucoma is associated with optic nerve head ischemia. Several studies indicate that a disturbed autoregulation might contribute to glaucomatous optic neuropathy. Currently, five classes of intraocular pressure (IOP) reducing drugs are available for topical therapy in patients with glaucoma or elevated intraocular pressure. These drugs have also vasoactive properties, which may influence both the resting ocular circulation and the autoregulatory mechanisms of blood flow during changes in ocular perfusion pressure.

Study objective

To investigate the influence of common topical glaucoma therapy on ONH blood flow regulation during changes in IOP and systemic arterial blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 1 Dpt.

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Presence of intraocular pathology: ocular hypertension, glaucoma, retinal vasculopathy or other retinal diseases

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Ocular perfusion pressure - ONH blood flow relationship | on 2 study days

SECONDARY OUTCOMES:
Composite measure: Blood pressure, heart rate | on 2 study days

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Fuchsjaeger-Mayrl, MD, Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria